CLINICAL TRIAL: NCT07186855
Title: The Study on the Relationship Between Perioperative and Postoperative Circulating Tumor Cell Monitoring and Prognosis in Patients With Non-Small Cell Lung Cancer at Different Stages
Brief Title: Perioperative and Postoperative Circulating Tumor Cell Monitoring in Different Stage of NSCLC
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: LC2020L02
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early-stage NSCLC: CTC detection will be conducted on 180 cases.
  Interventions: Other: Blood Sample Collection for CTC Detection
- Advanced-Stage Non-Small Cell Lung Cancer: CTC detection will be conducted on 320 cases.
  Interventions: Other: Blood Sample Collection for CTC Detection

INTERVENTIONS:
Other: Blood Sample Collection for CTC Detection — Blood Sample Collection for CTC Detection

SUMMARY:
The study aims to enroll 500 non-small cell lung cancer patients at various stages and to employ this technology for CTC detection, with subsequent cytomorphological and chromosomal analysis of the isolated CTCs, and comprehensively assess the utility of this CTC monitoring technology in predicting postoperative recurrence, metastasis, and survival in non-small cell lung cancer patients across different stages.

DETAILED DESCRIPTION:
Lung cancer currently has the highest incidence and mortality rates among malignant tumors in China. Distant metastasis is one of the main causes of death in lung cancer patients, with hematogenous dissemination being the primary pathway for lung cancer metastasis. Theoretically, even at the carcinoma in situ stage, cancer cells can disseminate into the peripheral blood, forming circulating tumor cells (CTCs), thus playing a critical role in the process of distant metastasis in lung cancer. Early diagnosis and monitoring of recurrence and metastasis are essential for improving patient survival rates. Traditional methods for monitoring postoperative recurrence and metastasis in lung cancer patients rely primarily on imaging studies; however, by the time recurrence or metastasis is detected through imaging, the disease is often at an advanced stage, leading to suboptimal treatment outcomes. Previous studies have shown that changes in CTC levels usually precede the appearance of detectable lesions on imaging. Therefore, CTC level monitoring can predict recurrence, metastasis, treatment response, and prognosis in lung cancer patients.

As a form of "liquid biopsy," CTC testing can provide timely insights into a patient's disease status and offer better individualized treatment strategies for lung cancer patients. This study utilizes the viral tracing method developed by our research team, which holds independent intellectual property rights, as the primary technology. In addition, microfluidic technology has been introduced upstream in the workflow to initially screen and enrich CTCs, followed by ex vivo identification and characterization of the captured CTCs. The study aims to enroll 500 non-small cell lung cancer patients at various stages and to employ this technology for CTC detection, with subsequent cytomorphological and chromosomal analysis of the isolated CTCs. Finally, by integrating preoperative and postoperative imaging data, pathological findings, and recurrence, metastasis, and survival outcomes, we will comprehensively assess the utility of this CTC monitoring technology in predicting postoperative recurrence, metastasis, and survival in non-small cell lung cancer patients across different stages.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age of the patient: ≥18 and ≤75 years; (2) No prior anticancer treatment before surgery; (3) No history of other tumors, past or concurrent; (4) Underwent radical surgery for lung cancer between November 2020 and October 2022; (5) Postoperative pathological diagnosis of non-small cell lung cancer, with staging between Ia and IIIb; (6) Able to comply with study requirements and has signed informed consent.

Exclusion Criteria:

* (1) Patients with non-small cell lung cancer who have received tumor-related treatments before surgery (including chemotherapy, radiotherapy, targeted therapy, and immunotherapy); (2) Patients with severe cardiac, pulmonary, hepatic, cerebral, or renal dysfunction who are unable to tolerate surgery; (3) Pregnant patients; (4) Patients with concurrent other malignancies; (5) Patients with severe underlying diseases that make them unable to tolerate surgery; (6) Patients with types of lung cancer other than non-small cell lung cancer or with secondary malignant tumors in the lung.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 500 non-small cell lung cancer patients undergoing surgical treatment will be enrolled from the Department of Thoracic Surgery at the Cancer Hospital, Chinese Academy of Medical Sciences, and its affiliated centers.Among them, approximately 180 cases will be early-stage.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Two-Year Recurrence Status | Up to 2 years after surgery
  Time from surgery util recurrence

CONTACTS AND LOCATIONS:
Overall Officials: YOUSHAN MAO, MD, Study Director — NCC, CICAMS
Locations (1):
- Nationa Cancer Center, National Clinical Research Center for Cancer, Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijingn, China

IPD SHARING:
Plan to Share IPD: No
In accordance with relevant laws and regulations, researchers who wish to access the raw data should contact the principal investigator via email.